CLINICAL TRIAL: NCT03681717
Title: A Pragmatic Randomized Controlled Trial of Virtual Reality vs. Standard-of-Care for Comfort During Laceration Repair
Brief Title: Virtual Reality vs. Standard-of-Care for Comfort During Laceration Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Doctors of BC (Unknown)
Responsible Party: Principal Investigator, Ran Goldman, Professor and Co-head of the Division of Clinical Pharmacology, Division of Emergency Medicine, Department of Pediatrics; Investigator, BC Children's Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-02711
Record Dates: First submitted 2018-07-05; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Laceration
Keywords: Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Lacerations; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants are distracted by wearing the virtual reality headset and watching a roller coaster app during laceration repair with sutures.
  Interventions: Device: Virtual Reality
- Control (Standard-of-Care) (No Intervention): Participants are distracted with Standard-of-Care by doctors, nurses, nurse practitioners, child life specialists and/or parents.

INTERVENTIONS:
Device: Virtual Reality — Participants wear a Virtual Reality headset that consists of a ASUS phone and a ReTrack Utopia 360 VR Headset. The phone runs the VR Roller Coaster app to produce the virtual environment.
  Arms: Virtual Reality

SUMMARY:
Lacerations are a common reason for presentation to the Emergency Department and children needing laceration repair with sutures are experiencing pain and anxiety.

Virtual Reality (VR) is an immersive experience using sight, sound, and position sense. Using VR may enhance distraction during the painful procedure and may reduce attention to pain.

This study will randomize children (6 - 16 years old) to receive Virtual Reality or standard of care in addition to pharmacoanalgesia during a laceration repair procedure. Investigators will measure pain, anxiety, satisfaction, amount of analgesia and the length of procedure and compare between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 - <17 years
* Arriving to the Emergency Department with a chief complaint of laceration
* The managing physician determines need for repair with suture
* Parents will sign a consent form and children will sign an assent form

Exclusion Criteria:

* Children with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay)
* Triage category 1 (resuscitation)
* Facial features or injury prohibiting wearing VR goggles

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain using the Faces Pain Scale - Revised. | Pain is reported by children immediately following completion of the laceration repair
  Level of pain as reported by children using Faces Pain Scale - Revised. The scale includes six faces that represent progressively more intense features of pain. Children point to the face that best represents their current level of pain. The minimum score is 0 (representing least pain) and the maximum score is 10 (representing greater pain). The scale increase in increments of 2.

SECONDARY OUTCOMES:
Anxiety using the Venham Situational Anxiety Score | Anxiety is reported by children immediately following completion of the laceration repair
  Level of Situational Anxiety as reported by children using the Venham Situational Anxiety Score. This scale includes 8 sets of 2 images of children which represent differing levels of anxiety. Children point to the child that best represents them in that instance. In each set of 2 images of children, one represents greater anxiety (scored as 1) and one represents lesser anxiety (scored as 0). The points from each set of images are totaled. The minimum score is 0 (least anxious) and maximum score is 8 (most anxious).
Patient Satisfaction determined qualitatively by an open ended question | Satisfaction question is reported by children immediately following completion of the laceration repair
  Satisfaction from the procedure is determined qualitatively. Children are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).
Parent Satisfaction determined qualitatively by an open ended question | Satisfaction question is reported by parents immediately following completion of the laceration repair
  Satisfaction from the procedure is determined qualitatively. Parents are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).
Medication Dose | These will be recorded during the procedure and immediately following the procedure using the patient chart and nursing notes
  How much topical or local anesthetics are used and when they are used (24 hour time); how much sedatives are used and when they are used (24 hour time); how much analgesics are used and when they are used (24 hour time).
Timing | Documented immediately after patient and family given discharge paperwork
  Time in minutes from readiness for procedure (availability of child, staff and equipment) until completion of procedure (physician does not need to touch the patient anymore) and until discharged from the emergency department (given discharge paperwork).

CONTACTS AND LOCATIONS:
Overall Officials: Ran D. Goldman, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No